CLINICAL TRIAL: NCT06468410
Title: The Influence of Hatha Yoga Duration on Pulmonary Function in Sedentary Youth: An Acute and Four-Week Intervention Study
Brief Title: Effect of Hatha Yoga on Pulmonary Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monira Aldhahi (Other)
Collaborators: Çankırı Karatekin University (Other); Bandırma Onyedi Eylül University (Other)
Responsible Party: Sponsor-Investigator, Monira Aldhahi, Associate professor, Princess Nourah Bint Abdulrahman University
Organization: Princess Nourah Bint Abdulrahman University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-34
Record Dates: First submitted 2024-06-12; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: pulmonary function; yoga; students; exercise duration
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three groups:
  1. 60-minute Hatha Yoga group (60mHY, n=21)
  2. 30-minute Hatha Yoga group (30mHY, n=21)
  3. Control group (CG, n=21)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 60-minute Hatha Yoga group (Active Comparator): • 60mHY Group: Participants will undergo a 60-minute hatha yoga session twice a week for four weeks.
  Interventions: Other: short duration Hatha Yoga
- 30-minute Hatha Yoga group (Active Comparator): • 30mHY Group: Participants will undergo a 30-minute hatha yoga session twice a week for four weeks.
  Interventions: Other: long duration Hatha Yoga
- Control group (Placebo Comparator): • Control Group: Participants will receive information about physical activity guidelines but will not engage in any structured yoga exercise during the study period.
  Interventions: Other: Control group

INTERVENTIONS:
Other: long duration Hatha Yoga — 60 min of Hatha yoga for 4 weeks. Week One:Participants begin with foundational breathing and yoga practicesOn the second day, Square Breathwork is introduced to foster calm and concentration. After a warm-up, the yoga flow focuses on heart openers to increase chest and shoulder flexibility, ending with a soothing cool-down. Week Two:Advanced breathing techniques and targeted yoga flows are introduced. The second session includes Nadi Shodhana to balance the nervous system. Week Three:The focus remains on heart openers with varied breathing exercises. The second day revisits Full Yogic Breath, followed by a warm-up and another heart opener sequence, concluding with a cool-down. Week Four:The final week integrates additional breathing techniques. The last session features Kapalabhati and Suddhi Pranayama to purify and energize the body. After a warm-up, participants engage in a well-rounded yoga flow combining various poses to enhance overall fitness, concluding with a final cool-down.
  Arms: 30-minute Hatha Yoga group
Other: short duration Hatha Yoga — 30 min of Hatha yoga for 4 weeks .
  Arms: 60-minute Hatha Yoga group
Other: Control group — participants will receive information about physical activity guidelines but will not engage in any structured yoga exercise during the study period.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to to investigate the acute and chronic effects of a four-week hatha yoga (HY) exercise program with different durations (60 min and 30 min) on pulmonary function in sedentary young individuals.. The main questions it aims to answer are:

• Does a four-week hatha yoga (HY) more effective than 30 min of a four-week hatha yoga (HY) and the control group in improving the pulmonary function? Researchers will compare a four-week OF 60 min duration hatha yoga (HY) , 30 min duration of HY and control to see the differences in the pulmonary function among high school sedentary students

Participants will:

Participants will be randomly assigned to one of three groups:

1. 60-minute Hatha Yoga group (60mHY, n=21)
2. 30-minute Hatha Yoga group (30mHY, n=21)
3. Control group (CG, n=21)

DETAILED DESCRIPTION:
Objective: To investigate the acute and chronic effects of a four-week hatha yoga (HY) exercise program with different durations (60 minutes and 30 minutes) on pulmonary function in sedentary young individuals aged 15-16 years.

Study Design: Randomized Controlled Trial (RCT)

Participants:

• Sample Size: 52 sedentary individuals

Inclusion Criteria:

* High school adolescence
* Showed Sedentary lifestyle (defined as not participating in regular physical activity for at least 6 months.

Exclusion Criteria:

* Any known history of pulmonary, cardiovascular, or musculoskeletal conditions that would contraindicate exercise,
* participation in any other exercise program during the study period
* obesity (BMI > 25.00)
* Participants who are in medication that stimulate the heart of medication such as antibiotic use were excluded from the study

Randomization:

Participants will be randomly assigned to one of three groups:

4. 60-minute Hatha Yoga group (60mHY, n=21) 5. 30-minute Hatha Yoga group (30mHY, n=21) 6. Control group (CG, n=21)

Intervention:

* 60mHY Group: Participants will undergo a 60-minute hatha yoga session twice a week for four weeks.
* 30mHY Group: Participants will undergo a 30-minute hatha yoga session twice a week for four weeks.
* Control Group: Participants will receive information about physical activity guidelines but will not engage in any structured yoga exercise during the study period.

Outcome Measures:

• Primary Outcome: Pulmonary function measured by spirometry.

ELIGIBILITY:
Inclusion Criteria:

* High school adolescence
* Sedentary lifestyle (defined as not participating in regular physical activity for at least 6 months.

Exclusion Criteria:

* Any known history of pulmonary, cardiovascular, or musculoskeletal conditions that would contraindicate exercise,
* participation in any other exercise program during the study period
* obesity (BMI > 25)
* Participants who are on medication that stimulates the heart of medication such as antibiotic use were excluded from the study

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | at baseline and end of 4 week
  the maximum amount of air a person can exhale after taking a deep breath measured using spirometry
Forced Expiratory Volume in 1 second (FEV1) | at baseline and end of 4 week
  spirometry will be used to measure Forced Expiratory Volume in 1 second (FEV1). It is the volume of air (in liters) exhaled in the first second during forced exhalation after maximal inspiration.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Soyler, Phd, Principal Investigator — Bandırma Onyedi Eylül University
Locations (1):
- Bandirma Onyedi Eylul University, Balıkesir, Turkey (Türkiye)